CLINICAL TRIAL: NCT02152956
Title: A Phase 1/2, First in Human, Dose Escalation Study of MGD006, a CD123 x CD3 DART® Bi-Specific Antibody Based Molecule, in Patients With Relapsed or Refractory AML or Intermediate-2/High Risk Myelodysplastic Syndrome (MDS)
Brief Title: Flotetuzumab in Primary Induction Failure (PIF) or Early Relapse (ER) Acute Myeloid Leukemia (AML)
Acronym: VOYAGE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGD006-01
Expanded Access: NCT04678466 (No longer available)
Record Dates: First submitted 2014-05-28; First posted 2014-06-02 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: AML
Keywords: AML; leukemia; myelogenous; myeloid; refractory
MeSH Terms: conditions — Leukemia | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Cohort 0-a (Experimental)
  Interventions: Biological: Flotetuzumab 3 ng/kg/day, 4 days on and 3 days off
- Cohort 0-b (Experimental)
  Interventions: Biological: Flotetuzumab 10 ng/kg/day, 4 days on and 3 days off
- Cohort 0-c (Experimental)
  Interventions: Biological: Flotetuzumab 30 ng/kg/day, 4 days on and 3 days off
- Cohort 0-d (Experimental)
  Interventions: Biological: Flotetuzumab 100 ng/kg/day, 4 days on and 3 days off
- Cohort 1 (Experimental)
  Interventions: Biological: Flotetuzumab 300 ng/kg/day, 4 days on 3 days off, after one-step lead-in dose
- Cohort 2 (Experimental)
  Interventions: Biological: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after one-step lead-in dose
- Cohort 2a (Experimental)
  Interventions: Biological: Flotetuzumab 500 ng/kg/day, continuous infusion, after multi-step lead-in dose
- Cohort 3 (Experimental)
  Interventions: Biological: Flotetuzumab 700 ng/kg/day, 4 days on 3 days off, after multi-step lead-in dose
- Cohort 6 (Experimental)
  Interventions: Biological: Flotetuzumab 300 ng/kg/day, continuous infusion, after multi-step lead-in dose
- Cohort 7 (Experimental)
  Interventions: Biological: Flotetuzumab 500 ng/kg/day, continuous infusion, after multi-step lead-in dose
- Cohort 8 (Experimental)
  Interventions: Biological: Flotetuzumab 700 ng/kg/day, continuous infusion, after multi-step lead-in dose
- MTD Expansion (Experimental)
  Interventions: Biological: Flotetuzumab 500 ng/kg/day, continuous infusion, after multi-step lead-in dose
- MTD expansion with Ruxolitinib (Experimental)
  Interventions: Biological: Flotetuzumab 500 ng/kg/day, continuous infusion, after multi-step lead-in dose; Drug: Ruxolitinib

INTERVENTIONS:
Biological: Flotetuzumab 3 ng/kg/day, 4 days on and 3 days off — Flotetuzumab is a CD123 x CD3 bispecific antibody-based molecular construct referred to as a DART® molecule.
  Other Names: MGD006
  Arms: Cohort 0-a
Biological: Flotetuzumab 10 ng/kg/day, 4 days on and 3 days off — Flotetuzumab is a CD123 x CD3 bispecific antibody-based molecular construct referred to as a DART molecule.
  Other Names: MGD006
  Arms: Cohort 0-b
Biological: Flotetuzumab 30 ng/kg/day, 4 days on and 3 days off — Flotetuzumab is a CD123 x CD3 bispecific antibody-based molecular construct referred to as a DART molecule.
  Other Names: MGD006
  Arms: Cohort 0-c
Biological: Flotetuzumab 100 ng/kg/day, 4 days on and 3 days off — Flotetuzumab is a CD123 x CD3 bispecific antibody-based molecular construct referred to as a DART molecule.
  Other Names: MGD006
  Arms: Cohort 0-d
Biological: Flotetuzumab 300 ng/kg/day, 4 days on 3 days off, after one-step lead-in dose — Flotetuzumab is a CD123 x CD3 bispecific antibody-based molecular construct referred to as a DART molecule.
  Other Names: MGD006
  Arms: Cohort 1
Biological: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after one-step lead-in dose — Flotetuzumab is a CD123 x CD3 bispecific antibody-based molecular construct referred to as a DART® molecule.
  Other Names: MGD006
  Arms: Cohort 2
Biological: Flotetuzumab 500 ng/kg/day, continuous infusion, after multi-step lead-in dose — Flotetuzumab is a CD123 x CD3 bispecific antibody-based molecular construct referred to as a DART molecule.
  Other Names: MGD006
  Arms: Cohort 2a; Cohort 7; MTD Expansion; MTD expansion with Ruxolitinib
Biological: Flotetuzumab 700 ng/kg/day, 4 days on 3 days off, after multi-step lead-in dose — Flotetuzumab is a CD123 x CD3 bispecific antibody-based molecular construct referred to as a DART molecule.
  Other Names: MGD006
  Arms: Cohort 3
Biological: Flotetuzumab 700 ng/kg/day, continuous infusion, after multi-step lead-in dose — Flotetuzumab is a CD123 x CD3 bispecific antibody-based molecular construct referred to as a DART molecule.
  Other Names: MGD006
  Arms: Cohort 8
Drug: Ruxolitinib — Oral inhibitor of JAK kinase
  Other Names: Jakafi
  Arms: MTD expansion with Ruxolitinib
Biological: Flotetuzumab 300 ng/kg/day, continuous infusion, after multi-step lead-in dose — Flotetuzumab is a CD123 x CD3 bispecific antibody-based molecular construct referred to as a DART molecule.
  Arms: Cohort 6

SUMMARY:
Open-label, multi-dose, single-arm, multi-center, Phase 1/2 study conducted in three segments: the Single Patient Dose Escalation Segment (complete), followed by the Multi-Patient Dose Escalation Segment (complete) and the Maximum Tolerated Dose and Schedule (MTDS) Expansion Cohort Segment (closed). Having characterized safety and determined the maximum tolerated dose and schedule, the primary objective of this study now is to assess the anti-neoplastic activity of flotetuzumab in patients with PIF/ER AML, as determined by the proportion of patients who achieve CR or CRh. Starting with Cycle 2, patients who are benefiting from flotetuzumab may receive up to a maximum of 8 cycles of treatment.

Patients will receive daily increasing doses of flotetuzumab for the first week of Cycle 1 (Lead-In Dosing) followed by 3 weeks of continuous intravenous infusion at a the assigned dose. Subsequent cycles are each 4 weeks of continuous infusion at the assigned dose. Dosing may continue for up to 8 cycles. Follow up visits may continue for 6 months after treatment is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary or secondary AML [any subtype except acute promyelocytic leukemia (APL)] according to World Health Organization (WHO) classification
* Patients with AML must meet one of the following criteria, a or b:

  1. Primary Induction Failure (PIF) AML, defined as disease refractory to either, i or ii:

     * i. An intensive induction attempt, per institution. Induction attempts include high-dose and/or standard-dose cytarabine ± an anthracyclines/anthracenedione ± an anti-metabolite, with or without growth factor or targeted therapy containing regimens. Examples include but are not limited to: 1 cycle of high dose cytarabine (HiDAC) containing regimen, 1 cycle of liposomal cytarabine and daunorubicin, 2 cycles of standard dose cytarabine containing regimen
     * ii. For adults who are age 75 years or older, or who have comorbidities that preclude use of intensive induction chemotherapy; PIF is defined as AML refractory to one of the following less intensive regimens: i ≥ 2 but ≤ 4 cycles of Bcl-2 inhibitors in combination with azacitidine, decitabine, or low dose cytarabine, or ii ≥ 2 but ≤ 4 cycles of gemtuzumab ozogamicin monotherapy
  2. Early relapse (ER) AML, defined as AML in first relapse with initial CR1 duration < 6 months
* Limit of 3 prior lines of therapy (excluding focal radiation therapy for palliative purposes): up to 2 induction (induction, re-induction) or 1 induction plus/minus 1 consolidation attempt, followed by a maximum of 1 salvage/re-induction attempt.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Life expectancy of at least 4 weeks
* Peripheral blast count </= 20,000/mm3 at the time of first dose
* Acceptable laboratory parameters and adequate organ reserve

Exclusion Criteria:

* History of allogeneic stem cell transplantation
* Prior treatment with an anti-CD123-directed agent
* Need for concurrent other cytoreductive chemotherapy
* Any active untreated autoimmune disorders (with the exception of vitiligo, resolved childhood atopic dermatitis, prior Grave's disease now euthyroid clinically and with stable supplementation)
* Second primary malignancy that requires active therapy. Adjuvant hormonal therapy is allowed.
* Antitumor therapy or investigational agent within 14 days or 5 half-lives of Cycle 1 Day 1.
* Requirement, at the time of study entry, for concurrent steroids > 10 mg/day of oral prednisone or the equivalent, except steroid inhaler, otic preparations, nasal spray or ophthalmic solution
* Use of immunosuppressant medications in the 2 weeks prior to Cycle 1 Day 1
* Use of granulocyte colony stimulating or granulocyte-macrophage colony stimulating factor in the 2 weeks prior to Cycle 1 Day 1
* Known central nervous system (CNS) leukemia
* Active uncontrolled infection (including, but not limited to viral, bacterial, fungal, or mycobacterial infection),
* Known human immunodeficiency virus infection, unless all of the following criteria are met: CD4+ count ≥ 350 cells/μL, undetectable viral load, and receiving highly active antiretroviral therapy.
* Known, active, history of or current acute or chronic hepatitis B or C virus (HBV) infection (as evidenced by detectable HBV surface antigen and HBV DNA ≥ 500 IU/mL),
* History of hepatitis C virus (HCV) infection, unless the infection has been treated and cured,
* Active SARS-CoV-2 infection. While SARS-CoV-2 testing is not mandatory for study entry, testing for ongoing infection should follow local clinical practice guidelines/standards. Participants with a positive test result for ongoing SARS-CoV-2 infection, known asymptomatic infection, or suspected infection are excluded unless or until asymptomatic and with subsequent negative SARS-CoV-2 laboratory test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2014-06-09 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley L. Ward, MD, Study Director — MacroGenics
Locations (43):
- United States (20):
  - City of Hope National Medical Center, Duarte, California
  - UCSD Moores Cancer Center, La Jolla, California
  - UCSF - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Georgetown University - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Loyola University Chicago - Cardinal Bernadin Cancer Center, Maywood, Illinois
  - University of Maryland, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Stony Brook Medicine, Stony Brook, New York
  - University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (4):
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Institut Universitaire du Cancer de Toulouse-Oncopole, Toulouse
  - CHRU de Tours - Hôpital Bretonneau, Tours
- Germany (7):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinik Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - III. Med. Klinik-Klinikum rechts der Isar-Technische Universität München, Munich
  - Medizinische Klinik und II, Universitätsklinikum Würzburg, Würzbur
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
- Italy (4):
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola
  - University Vita-Salute San Raffaele, Milan
  - Unità Operativa di Ematologia Ospedale Santa Maria delle Croci, Ravenna
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Erasmus University Medical Center, Rotterdam
- Spain (2):
  - Universitat Autonomaa de Barcelona (UAB) - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - King's Health Partners, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Uy GL, Aldoss I, Foster MC, Sayre PH, Wieduwilt MJ, Advani AS, Godwin JE, Arellano ML, Sweet KL, Emadi A, Ravandi F, Erba HP, Byrne M, Michaelis L, Topp MS, Vey N, Ciceri F, Carrabba MG, Paolini S, Huls GA, Jongen-Lavrencic M, Wermke M, Chevallier P, Gyan E, Recher C, Stiff PJ, Pettit KM, Lowenberg B, Church SE, Anderson E, Vadakekolathu J, Santaguida M, Rettig MP, Muth J, Curtis T, Fehr E, Guo K, Zhao J, Bakkacha O, Jacobs K, Tran K, Kaminker P, Kostova M, Bonvini E, Walter RB, Davidson-Moncada JK, Rutella S, DiPersio JF. Flotetuzumab as salvage immunotherapy for refractory acute myeloid leukemia. Blood. 2021 Feb 11;137(6):751-762. doi: 10.1182/blood.2020007732. PMID 32929488

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 0-a: Flotetuzumab 3 ng/kg/day, 4 days on and 3 days off
- Cohort 0-b: Flotetuzumab 10 ng/kg/day, 4 days on and 3 days off
- Cohort 0-c: Flotetuzumab 30 ng/kg/day, 4 days on and 3 days off
- Cohort 0-d: Flotetuzumab 100 ng/kg/day, 4 days on and 3 days off
- Cohort 1: Flotetuzumab 300 ng/kg/day, 4 days on 3 days off, after lead-in dose
- Cohort 2: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after one-step lead-in dose:
- Cohort 2a: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after multi-step lead-in dose
- Cohort 3: Flotetuzumab 700 ng/kg/day, 4 days on 3 days off, after lead-in dose:
- Cohort 6: Flotetuzumab 300 ng/kg/day, continuous infusion, after multistep lead-in dose
- Cohort 7; MTD Expansion: Flotetuzumab 500 ng/kg/day, continuous infusion, after multistep lead-in dose
- Cohort 8: Flotetuzumab 700 ng/kg/day, continuous infusion, after multistep lead-in dose
- MTD Expansion With Ruxolitinib: Flotetuzumab 500 ng/kg/day, continuous infusion, after multistep lead-in dose Ruxolitinib: Oral inhibitor of JAK kinase
Period: Overall Study
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Started | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 4 | 4 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Death | 0 | 3 | 3 | 4 | 1 | 2 | 6 | 6 | 4 | 5 | 3 | 143 | 12
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 4 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 0
Not completed — progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after lead-in dose
- Cohort 2a: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after multistep lead-in dose
- Cohort 3: Flotetuzumab 700 ng/kg/day, 4 days on 3 days off, after multistep lead-in dose
- Total: Total of all reporting groups
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib | Total
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (NA) — There is only 1 participant in cohort.0-a. Standard deviation is not applicable | 59.3 (21.28) | 56.4 (17.10) | 71.8 (16.54) | 58.3 (14.50) | 67.3 (11.64) | 53.0 (11.33) | 73.5 (5.92) | 64.0 (10.81) | 61.2 (20.17) | 70.0 (8.19) | 58.3 (14.29) | 65.7 (12.02) | 59.5 (14.36)
Age, Customized [Count of Participants; unit: Participants]
  18 - 65 | 1 | 3 | 3 | 1 | 2 | 2 | 5 | 1 | 3 | 2 | 1 | 121 | 6 | 151
  66 - 75 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 2 | 2 | 2 | 1 | 53 | 3 | 69
  >75 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 11 | 3 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 4 | 0 | 0 | 4 | 3 | 2 | 2 | 0 | 85 | 4 | 109
  Male | 1 | 2 | 2 | 0 | 3 | 4 | 2 | 3 | 4 | 3 | 3 | 100 | 8 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 15
  Not Hispanic or Latino | 1 | 3 | 5 | 4 | 3 | 2 | 6 | 6 | 6 | 5 | 2 | 145 | 12 | 200
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 25 | 0 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 12
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 14 | 3 | 22
  White | 1 | 4 | 5 | 3 | 3 | 3 | 4 | 6 | 4 | 5 | 3 | 133 | 9 | 183
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0 | 21
  Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 6
Region of Enrollment [Number; unit: participants]
  Netherlands | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 0 | 10
  United States | 1 | 4 | 5 | 4 | 3 | 4 | 4 | 4 | 5 | 3 | 1 | 120 | 12 | 170
  Italy | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 8 | 0 | 12
  United Kingdom | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5
  France | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 26 | 0 | 28
  Germany | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 15 | 0 | 17
  Spain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Based on CR or CRh Rate
Description: Proportion of patients achieving a best response of CR (morphologic CR [mCR], cytogenetic CR [CRc], molecular CR [CRm], or CRh per Interworking Group AML response criteria.
  CR is defined as mCR, CRc, CRm or CRh. mCR is defined as: normal. neutrophil and platelet counts, less than 5% blast cells in a bone marrow (BM) smear and. no extramedullary disease.
  CRc is defined as: CR with no evidence of cytogenetic abnormalities in the bone marrow.
  CRm is defined as: CR with no evidence of molecular abnormalities in the bone marrow.
  CRh is defined as: CR with partial hematologic recovery.
Time Frame: up to 14 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 7: Flotetuzumab 500 ng/kg/day, continuous infusion, after lead-in dose
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 16 | 4

2. Secondary Outcome: Overall Complete Response Rate
Description: Rate of CR + CRh + CRi (CR with incomplete blood cell recovery [CR with incomplete neutrophil {CRn}or platelet recovery {CRp}]) + MLFS (morphologic leukemia-free state)
Time Frame: up to 14 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Flotetuzumab 300 ng/kg/day, 4 days on 3 days off, after lead-in dose:
- Cohort 2: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after lead-in dose:
- Cohort 2a: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after multistep lead-in dose:
- Cohort 3: Flotetuzumab 700 ng/kg/day, 4 days on 3 days off, after multistep lead-in dose:
- Cohort 6: Flotetuzumab 300 ng/kg/day, continuous infusion, after multistep lead-in dose:
- Cohort 7; MTD Expansion: Flotetuzumab 500 ng/kg/day, continuous infusion, after multistep lead-in dose:
- Cohort 8: Flotetuzumab 700 ng/kg/day, continuous infusion, after multistep lead-in dose:
- MTD Expansion With Ruxolitinib: Flotetuzumab 500 ng/kg/day, continuous infusion, after multistep lead-in dose:
  Ruxolitinib: Oral inhibitor of JAK kinase
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 27 | 4

3. Secondary Outcome: CR Rate
Description: Proportion of patients achieving a best response of CR (morphologic CR [mCR], cytogenetic CR [CRc], or molecular CR [CRm] per Interworking Group AML response criteria.
  CR is defined as mCR, CRc, CRm or CRh. mCR is defined as: normal. neutrophil and platelet counts, less than 5% blast cells in a bone marrow (BM) smear and. no extramedullary disease.
  CRc is defined as: CR with no evidence of cytogenetic abnormalities in the bone marrow.
  CRm is defined as: CR with no evidence of molecular abnormalities in the bone marrow.
  CRh is defined as: CR with partial hematologic recovery.
Time Frame: up to 14 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2a: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after lead-in dose
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 13 | 2

4. Secondary Outcome: CRh Rate
Description: Proportion of patients achieving a best response of CRh per Interworking Group AML response criteria.
  CRh is defined as: CR with partial hematologic recovery.
Time Frame: up to 14 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Flotetuzumab 300 ng/kg/day, 4 days on 3 days off, after one-step lead-in dose
- Cohort 2: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after one-step lead-in dose
- Cohort 2a; Cohort 7; MTD Expansion: Flotetuzumab 500 ng/kg/day, continuous infusion, after multi-step lead-in dose
- Cohort 3: Flotetuzumab 700 ng/kg/day, 4 days on 3 days off, after multi-step lead-in dose
- Cohort 6: Flotetuzumab 300 ng/kg/day, continuous infusion, after multi-step lead-in dose
- Cohort 8: Flotetuzumab 700 ng/kg/day, continuous infusion, after multi-step lead-in dose
- MTD Expansion With Ruxolitinib: Flotetuzumab 500 ng/kg/day, continuous infusion, after multi-step lead-in dose Ruxolitinib: Oral inhibitor of JAK kinase
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 14 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2

5. Secondary Outcome: Overall Response Rate
Description: Proportion of patients achieving a best response of CR, CRh, CRi, MLFS or partial response per Interworking Group AML response criteria.
  CR is defined as mCR, CRc, CRm or CRh. mCR is defined as: normal. neutrophil and platelet counts, less than 5% blast cells in a bone marrow (BM) smear and. no extramedullary disease.
  CRc is defined as: CR with no evidence of cytogenetic abnormalities in the bone marrow.
  CRm is defined as: CR with no evidence of molecular abnormalities in the bone marrow.
  CRh is defined as: CR with partial hematologic recovery.
Time Frame: up to 14 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2a: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after lead-in dose: Flotetuzumab is a CD123 x CD3 bispecific antibody-based molecular construct referred to as a DART® molecule.
- Cohort 3: Flotetuzumab 700 ng/kg/day, 4 days on 3 days off, after lead-in dose
- Cohort 6: Flotetuzumab 300 ng/kg/day, continuous infusion, after lead-in dose
- Cohort 8: Flotetuzumab 700 ng/kg/day, continuous infusion, after lead-in dose
- MTD Expansion: Flotetuzumab 500 ng/kg/day, continuous infusion, after lead-in dose
- MTD Expansion With Ruxolitinib: Flotetuzumab 500 ng/kg/day, continuous infusion, after lead-in dose Ruxolitinib: Oral inhibitor of JAK kinase
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 35 | 4

6. Secondary Outcome: HSCT Rate
Description: Rate of successful hematopoietic stem cell transplantation (HSCT) after the start flotetuzumab treatment and before subsequent therapy.
Time Frame: up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 1

7. Secondary Outcome: Occurrence of Dose Limiting Toxicity
Description: Maximum Tolerated Dose/Schedule: the MTDS is defined as the highest dose/schedule administered during any Cohort in the study at which the incidence of DLT is < 33% during the first cycle of MGD006 treatment.
Time Frame: Cycle 1 of a 28 day cycle.
Population: DLT were reported for dose escalation cohorts only (cohort 0-8)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 |  |

8. Secondary Outcome: Occurrence of Adverse Events (AEs)
Description: Cycle 1 through end of treatment
Time Frame: up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12

9. Secondary Outcome: Occurrence of Serious Adverse Events (SAEs)
Time Frame: up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 1 | 0 | 3 | 1 | 100 | 6

10. Secondary Outcome: Participants With Anti-drug Antibodies
Description: Occurrence of anti-drug antibody
Time Frame: Study Day 1, then every 28 days through 28-days after the last dose (up to 8 months)
Population: Participants were analyzed for the development of ADA regardless of dose level. Presence or absence of ADA is not related to dose level. The relevant information is the change from one status (positive, negative, or not tested) to a different status.
Measure: Count of Participants; unit: Participants
Groups:
- All Dose Levels: Participants were analyzed for the development of ADA regardless of dose level. Presence or absence of ADA is not related to dose level. The relevant information is the change from one status (positive, negative, or not tested) to a different status.
Arm/Group | All Dose Levels
Number analyzed (Participants) | 244
Participants
  Not tested at baseline, not tested on study | 144
  Not tested at baseline, all negative on study | 4
  Not tested at baseline, at least 1 positive on study | 0
  Negative at baseline, not tested on study | 25
  Negative at baseline, all negative on study | 70
  Negative at baseline, at least 1 positive on study | 1
  Positive at baseline, not tested on study | 0
  Positive at baseline, all negative on study | 0
  Positive at baseline, at least 1 positive on study | 0

11. Secondary Outcome: Number of Patients With Infusion Related Reaction (IRR)
Description: Determine safety and efficacy of tocilizumab in the treatment of IRR/CRS as measured by incidence of IRR/CRS
Time Frame: During study drug administration (up to 8 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 1 | 3 | 3 | 3 | 3 | 3 | 5 | 6 | 5 | 5 | 2 | 78 | 8

12. Secondary Outcome: Number of Patients With Cytokine Release Syndrome (CRS)
Time Frame: up to 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2a: Flotetuzumab 500 ng/kg/day, 4 days on 3 days off, after lead-in dose:
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 107 | 4

13. Secondary Outcome: Maximum Serum Concentration of Flotetuzumab
Description: Measure the pharmacokinetics (PK) of flotetuzumab
Time Frame: Study day 1, then every 28 days and 28 days after the last dose (up to 8 months)
Population: The PK analysis was conducted for patients receiving 10, 30, 100, 300, and 500 ng/kg/day. The study drug was administered as continuous IV dosing. Due to the short half-life, Cmax is not influenced by drug administration schedule. The data for all participants treated at a dose, regardless of schedule, were analyzed together. Specimens were collected and individually analyzed for concentrations only in the 700 ng/kg/day, no PK parameters were derived for this dose group.
Measure: Median (Full Range); unit: pg/mL
Groups:
- 10 ng/kg/Day: All patients treated at 10 mg/kg/day
- 30 ng/kg/Day: All patients treated at 30 mg/kg/day
- 100 ng/kg/Day: All patients treated at 100 mg/kg/day
- 300 ng/kg/Day: All patients treated at 300 mg/kg/day wither 4 days on/3 days off or by continuous infusion.
- 500 ng/kg/Day: All patients treated at 500 mg/kg/day wither 4 days on/3 days off or by continuous infusion.
Arm/Group | 10 ng/kg/Day | 30 ng/kg/Day | 100 ng/kg/Day | 300 ng/kg/Day | 500 ng/kg/Day
Number analyzed (Participants) | 4 | 5 | 4 | 9 | 212
pg/mL | 16.1 [5.55 to 25.3] | 34.5 [21.0 to 55.0] | 82.8 [68.2 to 180] | 177 [43.6 to 998] | 185 [51.8 to 754]

14. Secondary Outcome: Post-baseline Transfusion Independence Rate
Description: The number of patients who were transfusion-dependent at baseline and did not receive transfusions during any consecutive 56-day period will be calculated. The number of patients who are transfusion independent at baseline and remain independent during any 56-day post-baseline period will also be calculated.
Time Frame: 56 days
Population: No data was collected regarding transfusion dependency status at baseline or post-baseline.
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Patients Alive at 6 Months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 1 | 2 | 2 | 3 | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 42 | 6

16. Secondary Outcome: Event-free Survival
Description: Time from the first dose of study drug until date of evidence of primary refractory disease to flotetuzumab, relapse from CR, CRh or CRi, or death from any cause, whichever occurs first.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
months | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events.

17. Secondary Outcome: Mortality Rate
Description: number of deaths from any cause within 30, 60, 90, or 180 days of first dose of study drug
Time Frame: Throughout the study, up to 3 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants
  Mortality at 0-30 days | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 23 | 2
  Mortality at 31-60 days | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 34 | 3
  Mortality at 61-90 days | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 19 | 1
  Mortality at 91- >180 days | 1 | 2 | 2 | 4 | 0 | 1 | 4 | 4 | 4 | 2 | 1 | 67 | 6
  unknown | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 42 | 0

18. Secondary Outcome: Number of Patients Alive at 12 Months
Description: Number of patients alive at 1 year from first dose of study drug
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 4 | 3 | 6 | 6 | 6 | 5 | 3 | 185 | 12
Participants | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 16 | 3

19. Secondary Outcome: Median Time to Response
Description: Time from first dose of study drug to first CR, CRh, CRi, or MLFS
Time Frame: up to 14 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 6 | Cohort 3 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 43 | 6 | 6 | 6 | 5 | 3 | 185 | 12
months | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events. | NA [NA to NA] — Not estimable due to an insufficient number of participants with events.

20. Secondary Outcome: Duration of Response of Patients With CR or CRh
Description: Time of initial documentation of response to the time of disease relapse or death due to any cause, whichever occurs first.
Time Frame: Up to 2 years
Population: Analysis is based on the number of participants who had a CR or CRh as reported in Outcome Measure 1
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 16 | 4
Months |  |  |  |  |  |  |  | 4.0 (NA) — There was only 1 response in this cohort. |  | 2.3 (NA) — There was only 1 response in this cohort |  | 1.4 (1.04) | 1.1 (1.56)

21. Secondary Outcome: Overall Survival
Description: Time from first dose to death from any cause
Time Frame: Up to 2 years
Measure: Median (Standard Deviation); unit: months
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
Number analyzed (Participants) | 1 | 4 | 5 | 4 | 3 | 4 | 6 | 6 | 6 | 5 | 3 | 185 | 12
months | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events. | NA (NA) — Not estimable due to an insufficient number of participants with events.

22. Secondary Outcome: Rate of Hospitalization for Patients in the Expansion Cohort After Initial Discharge
Description: Initial dosing procedures were performed as a hospital inpatient. Incidence rate of hospitalization after discharge from the hospital will be calculated
Time Frame: up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | MTD Expansion
Number analyzed (Participants) | 185
Participants | NA — Not estimable due to an insufficient number of participants with events.

23. Secondary Outcome: Duration of Hospitalization for Patients in the Expansion Cohort
Description: Duration of hospitalization will be characterized after discharge from initial dosing will be characterized
Time Frame: up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | MTD Expansion
Number analyzed (Participants) | 185
Participants | NA — Not estimable due to an insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Throughout the study, up to 95 months.
Description: AEs are based on physical exam, patient reports, and significant abnormal laboratory values.
  AEs were not collected in survival follow up. Only SAEs were collected in survival follow up if related to study treatment.
  Only patients who received study treatments were assessed for safety. Progression of cancer causing hospitalization or death is not considered an SAE, unless considered drug-related by the investigator.[
Groups:
- MTD Expansion With Ruxolitinib: Flotetuzumab 500 ng/kg/day, continuous infusion, after lead-in dos Ruxolitinib: Oral inhibitor of JAK kinase
Arm/Group | Cohort 0-a | Cohort 0-b | Cohort 0-c | Cohort 0-d | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 3 | Cohort 6 | Cohort 7 | Cohort 8 | MTD Expansion | MTD Expansion With Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 0/1 | 3/4 | 3/5 | 4/4 | 2/3 | 2/4 | 6/6 | 6/6 | 5/6 | 5/5 | 3/3 | 144/185 | 12/12
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/4 | 0/5 | 2/4 | 1/3 | 2/4 | 2/6 | 1/6 | 0/6 | 3/5 | 1/3 | 100/185 | 6/12
Other Adverse Events (participants affected / at risk) | 1/1 | 4/4 | 5/5 | 4/4 | 3/3 | 4/4 | 6/6 | 6/6 | 6/6 | 5/5 | 3/3 | 185/185 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 0-a (N=1) | Cohort 0-b (N=4) | Cohort 0-c (N=5) | Cohort 0-d (N=4) | Cohort 1 (N=3) | Cohort 2 (N=4) | Cohort 2a (N=6) | Cohort 3 (N=6) | Cohort 6 (N=6) | Cohort 7 (N=5) | Cohort 8 (N=3) | MTD Expansion (N=185) | MTD Expansion With Ruxolitinib (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 12 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 7 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epstein-Barr viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scedosporium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 8 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronavirus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercapnic coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device infusion issue (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Central venous catheter removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 0-a (N=1) | Cohort 0-b (N=4) | Cohort 0-c (N=5) | Cohort 0-d (N=4) | Cohort 1 (N=3) | Cohort 2 (N=4) | Cohort 2a (N=6) | Cohort 3 (N=6) | Cohort 6 (N=6) | Cohort 7 (N=5) | Cohort 8 (N=3) | MTD Expansion (N=185) | MTD Expansion With Ruxolitinib (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 3 | 2 | 3 | 1 | 2 | 0 | 1 | 35 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 0 | 35 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 7 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 11 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 28 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 23 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 4 | 0 | 2 | 3 | 83 | 5
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 2 | 2 | 3 | 3 | 75 | 5
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 2 | 2 | 41 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 42 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 38 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 22 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 12 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 13 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 12 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 11 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 4 | 0 | 2 | 2 | 79 | 7
Fatigue (General disorders) | 0 | 2 | 2 | 1 | 1 | 1 | 2 | 2 | 4 | 0 | 0 | 43 | 1
Pyrexia (General disorders) | 0 | 0 | 2 | 2 | 2 | 0 | 3 | 3 | 2 | 2 | 2 | 37 | 4
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 16 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 15 | 2
Asthenia (General disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 7 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 95 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3 | 3 | 3 | 3 | 3 | 5 | 6 | 5 | 5 | 1 | 70 | 8
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 11 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 34 | 3
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 1 | 30 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 1 | 2 | 0 | 0 | 26 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 0 | 1 | 26 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 26 | 3
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 25 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 1 | 17 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 18 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 16 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 3 | 0 | 0 | 11 | 1
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 3 | 2 | 3 | 6 | 3 | 5 | 1 | 74 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 1 | 1 | 56 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 45 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 3 | 2 | 0 | 0 | 2 | 41 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 3 | 3 | 2 | 0 | 41 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 4 | 2 | 2 | 1 | 1 | 39 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 3 | 1 | 0 | 1 | 1 | 27 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 3 | 0 | 1 | 21 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 14 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 16 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 57 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 28 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 26 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 23 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 22 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 15 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 52 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 22 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 14 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 32 | 2
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 26 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 20 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 10 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 13 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 10 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 49 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 28 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 26 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 26 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 23 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 15 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 12 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 34 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 25 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 25 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 18 | 6
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 12 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 1 | 38 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 24 | 3
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 13 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT02152956/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT02152956/SAP_001.pdf